CLINICAL TRIAL: NCT03703544
Title: The Glycaemic Response of Local Foods Using the Continuous Glucose Monitoring System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Collaborators: Health Promotion Board, Singapore (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2017/00994
Record Dates: First submitted 2018-10-09; First posted 2018-10-12 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2019-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High glycemic index (Experimental): Subjects will consume locally consumed meals which are high glycemic index for breakfast, lunch snack and dinner will be provided.Participants' blood glucose will be monitored using the Continuous Glucose Monitor.
  Interventions: Other: High glycemic index
- Low glycemic index (Experimental): Subjects will consume locally consumed meals which are low glycemic index for breakfast, lunch snack and dinner will be provided. Participants' blood glucose will be monitored using the Continuous Glucose Monitor.
  Interventions: Other: Low glycemic index

INTERVENTIONS:
Other: High glycemic index — Wheat yellow noodle, glutinous rice, tea with sucrose, biscuits, jelly made with sucrose and teriyaki chicken rice.The foods provided have been tested as high glycemic index. Participants' blood glucose will be monitored using the Continuous Glucose Monitor.
  Arms: High glycemic index
Other: Low glycemic index — Beta-glucan yellow noodle, basmati rice, tea with isomaltulose, biscuits, jelly made with isomaltulose and mung bean noodles.The foods provided have been tested as low glycemic index.Participants' blood glucose will be monitored using the Continuous Glucose Monitor.
  Arms: Low glycemic index

SUMMARY:
This study is carried out to determine the effect of high and low GI of local foods using Continuous Glucose Monitoring System (CGMS™) on 24 hour blood glucose profiles.

DETAILED DESCRIPTION:
Glycemic Index (GI) is a method of classifying foods based on the food's ability to raise the blood glucose level. Low GI foods are recommended as Participants will have a lower impact on blood glucose concentrations. The research sets out to determine the effect of GI on 24 hour blood glucose profiles in healthy Chinese male participants. There will be two test sessions where participants will consume either a high or low GI breakfast, lunch, snack and dinner. Participants will take part in two test sessions (each spanning over 3 days and to monitor the participants' glycemic response using a Continuous Glucose Monitoring System (CGMS) throughout the period.This study specifically attempts to see how having high and low GI locally consumed meals impact on blood glucose.

ELIGIBILITY:
Inclusion Criteria:

* Chinese, male
* Age between 21-50 years
* Body mass index between 18 to 25 kg/m2
* Normal blood pressure (<140/90 Hgmm)
* Fasting blood glucose < 6 mmol/L

Exclusion Criteria:

* Current Smoker
* Have any metabolic diseases (such as diabetes, hypertension etc)
* Have known glucose-6-phosphate dehydrogenase deficiency (G6PD deficiency)
* have medical conditions and/or taking medications known to affect glycaemia (glucocorticoids, thyroid hormones, thiazide diuretics)
* Have an ongoing infection or currently undergoing treatment at the time of screening
* Known Chronic infection or known to suffer from or have previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV)• Have active Tuberculosis (TB) or currently receiving treatment for TB
* Have intolerances or allergies to any foods
* Partake in sports at the competitive and/or endurance levels

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male participants
Enrollment: 15 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
Daily blood glucose profile | 24 hours
  The daily total blood glucose response is measured for each low and high GI treatment as the area under the curve over 24 hours using CGMS for breakfast, lunch, snack and dinner.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No